CLINICAL TRIAL: NCT02489851
Title: Quadratus Lumborum Block vs Tranversus Abdominis Plane Block for Post Cesarean Section Analgesia. A Randomised Controlled Study
Brief Title: Quadratus Lumborum Block vs Tranversus Abdominis Plane Block for Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corniche Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ch23031404
Record Dates: First submitted 2015-07-02; First posted 2015-07-03 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2015-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quadratus Lumborum block group (Active Comparator): Quadratus Lumborum block group (QL)
  patients will receive a bilateral Quadratus Lumborum block using Bupivicaine 0.125%
  Interventions: Procedure: Quadratus Lumborum block
- Transversus abdominis plane block group (Active Comparator): Transversus abdominis plane block (TAP)
  patients will receive a bilateral TAP block using Bupivicaine 0.125%
  Interventions: Procedure: Tranversus Abdominis plane block

INTERVENTIONS:
Procedure: Quadratus Lumborum block — 0.2 ml/kg bupivicaine 0.125% injected bilateraly at the posterior border of the quadratus Lumborum muscle
  Other Names: QLB
  Arms: Quadratus Lumborum block group
Procedure: Tranversus Abdominis plane block — 0.2 ml/kg bupivicaine 0.125% injected bilateraly between internal oblique and transversus abdominis muscles.
  Other Names: TAP
  Arms: Transversus abdominis plane block group

SUMMARY:
The Quadratus Lumborum block (QLB) was first described by Blanco in 2007. The main advantage of QLB compared to the Transversus Abdominis Plane block (TAP) is the extension of local anesthetic agent beyond the TAP plane to the thoracic paravertebral space. The wider spread of the local anesthetic agents may produce extensive analgesia and prolonged action of the injected local anesthetic solution.

Previous studies showed that both TAP block and QLB may reduce morphine requirements in the postoperative period in patients who had cesarean section under spinal anaesthesia. However there are no published reports comparing the 2 techniques.

The aim of this randomised controlled, double blinded study is to compare the analgesic efficacy of QLB compared to TAP block in patients who had cesarean section under spinal anesthesia.

DETAILED DESCRIPTION:
After ethical committee approval, informed written consent will be obtained from all patients. A Sample size of 72 patients (36 per group) was calculated based on 15% reduction in morphine consumption with 0.05% significance and a power of 0.8.

Consenting patients scheduled to have elective cesarean section under spinal anesthesia will be randomised to receive bilateral QLB or TAP at the end of surgery.The dose of local anaesthetic in both groups will be 0.2 ml/kg 0.125% Bupivacaine. Allocation to either group will be done using closed envelope technique.

All the blocks will be performed in operation theatre after the end of cesarean section with intravenous access, ECG, BP, oxygen saturation by pulse oximetry monitoring and full resuscitation equipment and medication ready.

All patients will be in the supine position . Under ultrasound guidance a 22 Gauge, two inch Pajunk Sonoplex needle will be used for both techniques. The calculated dose of local anaeshetic will be injected bilateraly with intermittent aspiration. The spread of injectate will be seed on ultrasound.

All patients will receive the routine postoperative analgesia, comprising patient-controlled IV morphine analgesia and regular diclofenac and paracetamol.

All patients will be assessed postoperatively by a blinded investigator: in the postanesthesia care unit and at 2, 4, 6, 12, 24, 36, and 48 h postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Elective caesarean sections ASA 1 to 3 Written informed consent.

Exclusion Criteria:

Patient refusal Local infection at the site of injection Allergy to study medications Sepsis Anatomic abnormalities Systemic anticoagulation or coagulopathy Inability to comprehend or participate in pain scoring system Inability to use intravenous patient controlled analgesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Total morphine used in the first 48 hours after surgery | 48 hours
  Total cumulative morphine dose in mg used in the first 48 hours after surgery

SECONDARY OUTCOMES:
Severity of postoperative pain via visual analogue pain scale (VAS) | 48 hours
  VAS range from 0 for no pain to 10 for worst pain imaginable
Nausea or vomiting | 48 hours
  0 = No Nausea
  1. = Mild Nausea.
  2. = Moderate
  3. = Severe Nausea or Vomiting
Sedation score | 48 hours
  1. = drowsy but responds to normal verbal communication.
  2. = asleep, but awakes with verbal communication.
  3. = asleep, awakens with mild physical stimulation.
  4. = asleep, unresponsive to mild physical stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Rafa Blanco, FRCA, Principal Investigator — Corniche Hospital; Tarek Ansari, FFARCSI, Principal Investigator — Corniche Hospital; Nanda Shetty, MD, Principal Investigator — Corniche Hospital
Locations (1):
- Corniche Hospital, Abu Dhabi, United Arab Emirates

REFERENCES:
- [Derived] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488